CLINICAL TRIAL: NCT01207804
Title: A Single Center Feasibility Trial of the Safety and Efficacy of the ValenTx Endo Bypass System in Obese Patients
Brief Title: Feasibility Trial of ValenTx Endo Bypass System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ValenTx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIM
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental)
  Interventions: Device: ValenTx Endo Bypass System

INTERVENTIONS:
Device: ValenTx Endo Bypass System — Patient is implanted with device and followed for 12 weeks
  Other Names: ValenTx; Endo Bypass System; EBS

SUMMARY:
The purpose of the study is to provide initial clinical data to support the feasibility of use of the ValenTx Endo Bypass system in enhancing weight loss and co-morbidity resolution in morbidly obese patients.

DETAILED DESCRIPTION:
This is a single center open label feasibility study to evaluate the safety, efficacy and performance of the ValenTx Endo Bypass system.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age
* >=35 kg/m2 and <= 50 kg/m2, with or without comorbid conditions(s).
* Documented failure with non-surgical weight loss methods
* Willing to comply with study procedures and visit schedule
* Willing and able to provide Informed Consent

Exclusion Criteria:

* Pregnancy or intention of becoming pregnant within the study duration.
* Endoscopic lesions such as important hiatal hernia, gastric or duodenal ulcer, atresias or stenosis, polyps of the stomach.
* Subject with potential upper gastrointestinal bleeding such as esophageal or gastric varices, Mallory-Weis syndrome or congenital or acquired intestinal telangiectasia.
* Past history of esophageal or gastric/GI surgery, obstruction, adhesive peritonitis, or large hiatal hernia (> 3 cm).
* IBS, unexplained intermittent vomiting, severe abdominal pain or chronic constipation within 60 days of study day 1
* Unexplained anaemia, Pancreatitis, Portal hypertension, Esophagitis or Barrett's esophagus, known gallstones or anomalies of the GI tract
* Any bodily infections within 30 days of study day 1.
* Prolonged steroid use
* Hep C or HIV positive
* Known allergies to any of the device materials
* Use of weight loss medication or an investigational drug or device within 2 months prior to enrolment and throughout the study period.
* Recent or ongoing cancer, history of severe renal, hepatic, cardiovascular or pulmonary disease or transplants
* Inability to tolerate anti-inflammatory medications
* Evidence of psychiatric problems or dietary habits that would contraindicate study treatment;
* Active drug or alcohol addiction within 12 months of enrolment and throughout the study duration.
* Prior history of inflammatory diseases of the GI tract, (e.g., esophagitis, varices, gastric or duodenal ulceration, or Crohn's disease; congenital or acquired GI anomalies, e.g., bowel strictures)
* Ongoing treatment with anticoagulants, steroids, aspirin, NSAIDs, or other gastric irritants within 1 month prior to enrollment and throughout the study period.
* Participation in previous (within 60 days of study day 1) or ongoing clinical trial or current or past usage (within 60 days of study day 1) of investigation drug or device.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Device-related adverse events | 12 weeks

SECONDARY OUTCOMES:
Device performance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Rumbaut, MD, Principal Investigator — Hospital San Jose Tec
Locations (1):
- Hospital San Jose Tec de Monterrey, Monterrey, Mexico